CLINICAL TRIAL: NCT01653925
Title: Molecular Mechanisms of Dutasteride and Dietary Interventions to Prevent Prostate Cancer and Reduce Its Progression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: INAF-2010-H09-10-114
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prostatic Neoplasms; Low Grade Prostate Cancer
Keywords: Prostatic Neoplasms; Low grade prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary intervention first (Experimental): The dietary intervention will be aimed to increase intake of ω-3 long chain fatty acids and to reduce intake of saturated and trans fatty acids.
  Interventions: Other: Dietary intervention first
- Drug intervention first (Experimental): Intake of 5α-Reductase Inhibitor
  Interventions: Drug: Drug (Dutasteride) intervention first

INTERVENTIONS:
Other: Dietary intervention first — The dietary intervention will be aimed to increase intake of ω-3 long chain fatty acids and to reduce intake of saturated and trans fatty acids. Three consultations with a nutritionist experienced in clinical trials will be planned over a 6-month period. An additional 2 consultations in the last 6 months with the study nutritionist will be planned for men allocated to the dietary fat intervention arm first. Then, after the 6 months of diet intervention, drug intervention with 5α-Reductase Inhibitor will be add to diet for the 6 following months.
  Other Names: Dutasteride
  Arms: Dietary intervention first
Drug: Drug (Dutasteride) intervention first — 5α-Reductase Inhibitor will be taken daily in tablet dosage form (0.5 mg) taken orally for 12 months depend of the group. After 6 months of drug intake, dietary fat intervention will be add to treatment for the following 6 months. Three consultations with a nutritionist experienced in clinical trials will be planned over this 6-month period.
  Other Names: Dutasteride
  Arms: Drug intervention first

SUMMARY:
The purpose of this study is to determine whether marine omega-3 fatty acids and 5-alpha-reductase inhibitor are effective in the progression of prostate cancer for low-risk prostate cancer patients.

DETAILED DESCRIPTION:
The study has a duration of 1 year for each participant. Subjects will be first assigned to a dietary or a dutasteride intervention that they will consume for the first 6 months. After 6 months, all men will have a combined intervention of dutasteride and diet to complete follow-up of 12 months. This will allow us to study interactive effects.

Dietary intervention consists on a high w-3 long-chain fatty acids diet without supplement and to reduce intake of saturated and trans fatty acids.

Prostatic biopsies will be taken at time of diagnosis and at 6 and 12 months after the beginning of the study. Blood will be drawn before each prostate biopsy session and urine will be collected before each prostate biopsy and after digital rectal examination.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk prostatic neoplasms
* Candidate for active surveillance
* Informed consent

Exclusion Criteria:

* Current fish oil supplementation
* Current NSAID use

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10-28 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effects of the Interventions on Lipid Metabolism From Blood and Prostatic Microenvironment | 0-6-12 months
  In this aim the investigators will measure the effects of the interventions on the fatty acid profile of phospholipids from RBC and from snap frozen prostate tissue. Fatty acid profile from prostatic tissue has never been studied. The investigators aim that change in fatty acid intake will affect fatty acid profile of prostatic tissue. Fatty acid profile from red blood cells will serve as a marker of dietary fatty acid intake. Previous studies have shown that fatty acids profile from RBC differs from the one from muscle tissue and that the dietary effect on RBC fatty acids profile is almost maximal within 6 months.

SECONDARY OUTCOMES:
Effect of Interventions on Gene Expression Profile | 0-6-12 months
  In this aim the investigators will investigate how the interventions affect prostate tissue gene expression profile determined by cDNA micro-array analysis. We hypothesize that a down-regulation will occur in genes associated with inflammation, androgen synthesis, cell proliferation and angiogenesis pathways. Also, this prospective study provides an opportunity of a retrospective comparison of baseline gene expression patterns from initial prostate biopsy will be correlated with baseline self-reported dietary intake.
Effects of Interventions on Hormonal Metabolism | 0-6-12 months
  The investigators will initially focus our attention on estrogens (Estrone, Estradiol) and most important androgens and their metabolites (dihydrotestosterone, testosterone, 3-α-diolglucuronide, androsterone glucuronide).
Determine the Clinical Utility of Urine-Based Cancer Markers in the Context of Interventions to Reduce Cancer Progression | 0-6-12 months
  Although one of the best tumor markers available to monitor disease recurrence after treatment, PSA lacks specificity to monitor patients on active surveillance. The expression of urinary PCA3 (developed in Québec) improves the diagnosis of prostate cancer over standard parameters, including PSA, and the PCA3 score was shown to correlate with grade, stage and tumor volume in prostatectomy specimen. Another gene-based marker, the TMPRSS2-ERG gene fusion transcript, is also associated with tumor aggressiveness and detected in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Fradet, MD, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Hotel-Dieu of Quebec, Québec, Quebec
  - Institute of nutraceuticals and functional food of Laval University, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided